CLINICAL TRIAL: NCT04991402
Title: Obesogenic Origins of Maternal and Child Metabolic Health Involving Dolutegravir
Acronym: ORCHID
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Northwestern University (Other); University of Cape Town (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Hawaii (Other); Tufts University (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Senior Research Director, Columbia University
Other Study IDs: AAAT6112; 1R01HD104599 (NIH)
Record Dates: First submitted 2021-06-23; First posted 2021-08-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: HIV; Obesity; Obesity, Infant; Maternal Obesity During Childbirth; Maternal Obesity Complicating Pregnancy
Keywords: HIV; Dolutegravir; Metabolic health; Maternal obesity; Pregnancy
MeSH Terms: conditions — Obesity; Pediatric Obesity; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood, whole blood, plasma and serum, breastmilk, urine, adipose tissue (substudy participants only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Pregnant women living with HIV initiating Dolutegravir (DTG) in pregnancy (iDTG): Pregnant women living with HIV initiating DTG-based ART in pregnancy at the 1st visit
  Interventions: Device: Dolutegravir-based antiretroviral therapy
- Pregnant women living with HIV already on DTG-based ART prior to pregnancy (cDTG): Pregnant women living with HIV already on DTG-based ART prior to enrollment and continuing DTG use through pregnancy
  Interventions: Device: Dolutegravir-based antiretroviral therapy
- HIV uninfected pregnant women: Pregnant women not living with HIV

INTERVENTIONS:
Device: Dolutegravir-based antiretroviral therapy — This study focuses on the impact of Dolutegravir (DTG)-based antiretroviral therapy (ART) on metabolic health of women and children in pregnancy, delivery and beyond. In order to understand the potential adverse effects of DTG, pregnant women living with HIV- both those initialing DTG-based ART in pregnancy as well as those who were established on DTG-based ART prior to pregnancy, will be less than or equal to 18 weeks' gestation at enrollment to allow for detection of metabolic abnormalities as they begin to develop during the course of pregnancy.
  This is considered standard of care.
  Groups: Pregnant women living with HIV already on DTG-based ART prior to pregnancy (cDTG); Pregnant women living with HIV initiating Dolutegravir (DTG) in pregnancy (iDTG)

SUMMARY:
A total of 1900 pregnant women in the 1st trimester and their children will be enrolled and followed for two years (ORCHID study main cohort). As part of this, mother-infant pairs will be required to attend up to 10 study visits separate from routine clinic visits, these visits include 3 antenatal visits (less than or equal to 18, 24-28 and 32-36 weeks) and 16 postnatal visits (<2 and 6 weeks, 3, 6, 12, 18, and 24 months). Participants will also be asked to engage in long-term follow-up, with visits occurring every 6 months through Month 60 (at 30, 36, 42, 48, 54, and 60 months). Measurements in mothers will include demographics and health status, HIV disease and ART use, intercurrent medical history including concomitant medication use, HIV viral load testing, ART adherence, HIV antibody testing in women without HIV; body composition, caloric intake, dysglycemia and insulin resistance (IR), lipid profiles, anthropometry, resting energy expenditure, hepatic steatosis, specimen collection (whole blood, plasma, serum, urine, placenta and breastmilk), systemic and adipose inflammation, as well as metabolites, lipid subspecies and eicosanoids. Measurements in infants will include uterine gestational age and fetal growth, as well as metabolites, lipid subspecies and eicosanoids, body composition, dysglycemia and IR, lipid profiles, anthropometry, feeding, specimen collection (cord blood, whole blood, plasma and serum) and intercurrent medical history including concomitant medication use. Additional data on maternal health in pregnancy and birth outcomes will be abstracted from medical records.

DETAILED DESCRIPTION:
Dolutegravir (DTG)-based antiretroviral therapy (ART) is being scaled up as part of the preferred 1st-line ART regimen. However, DTG has recently been implicated as an obesogen that is associated with increased weight and adipose tissue gain compared to other antiretroviral agents. Obesity in pregnancy is associated with poor health outcomes for both mother and child as pregnancy is a critical period during which exposures leading to alterations in metabolic health may influence not only long-term maternal health but also fetal, neonatal, and ultimately child health. To address the gap of knowledge on the obesogenic effects of DTG in pregnant women living with HIV (WLHIV) and their children, this prospective cohort study will investigate the impact of DTG in pregnancy and its obesogenic effects on the metabolic health of WLHIV and their children, compared to women without HIV and their children. Up to 1900 pregnant women will be enrolled and followed to delivery and then as mother-infant pairs through 5 years postpartum (ORCHID study main cohort).

Additionally, a nested cohort study will be conducted and enroll a subset of 108 pregnant women who are currently being followed as part of the parent ORCHID study's main cohort. This substudy will explore the associations of DTG (initiating and continuing DTG use during pregnancy) with longitudinal perturbations in subcutaneous adipose tissue (SAT) function and changes in weight and adipose tissue mass in pregnancy through 2 years postpartum in WLHIV using a comparison group of HIV-seronegative women. They will been seen at up to 3 different time points (up to 2 visits during pregnancy and 1 visit postpartum) separate from the parent study to undergo a fat biopsy procedure to extract SAT samples.

ELIGIBILITY:
Inclusion Criteria:

For All Women:

* Confirmed pregnancy based on urine pregnancy test with viable gestation ≤ 18 weeks and 6 days by ultrasound
* Age 16 years or older
* No stated intention to relocate permanently outside of Cape Town through 2 years postpartum

For Women Living with HIV (WLHIV):

• Confirmed HIV infection based on medical record review and/or HIV antibody testing during antenatal care

For WLHIV continuing DTG in pregnancy (cDTG):

• Confirmed use of tenofovir 300mg + lamivudine 300mg/emtricitabine 200mg + dolutegravir 50mg (TLD) on the day of assessment

For WLHIV initiating DTG in pregnancy (iDTG):

• Planned initiation of TLD on the day of assessment or within 1 week thereafter, including women switching from efavirenz-based regimen

For women without HIV (HIV-):

• Confirmed HIV status by HIV antibody testing during antenatal care

Exclusion Criteria:

* In the opinion of the investigator, unable to provide informed consent due to mental or physical condition
* In the opinion of the investigator, unable to undertake BodPod assessment due to mental (eg, active psychosis or severe claustrophobia) or physical condition (eg, weight >250 kg).
* Currently being treated for any form of diabetes mellitus or hypertensive disorder based on participant self-report and medical record review

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants are pregnant women- some living with HIV and some HIV uninfected.
Study Population: The investigator will recruit up to 1900 pregnant women at their 1st antenatal clinic visit. Enrollment will be distributed across three main exposure categories by HIV status and Dolutegravir use: pregnant women living with HIV and initiating DTG-based ART in pregnancy (iDTG); pregnant women living with HIV already on DTG-based regimen prior to pregnancy and continuing DTG through pregnancy (cDTG); and pregnant women without HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 1920 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in excess gestational weight gain between pregnant women living with HIV and HIV negative pregnant women | <18 weeks (baseline), 32-34 weeks
  This is to measure the difference in gestational weight gain between pregnant women living with HIV and HIV negative pregnant women during pregnancy in kg. The women will be weighed by a scale at the study visit.
Difference in gestational weight gain between iDTG and cDTG pregnant women | <18 weeks (baseline), 32-34 weeks
  This is to measure the difference in gestational weight gain between pregnant women initiating DTG during pregnancy (iDTG) and pregnant women continuing DTG during pregnancy (cDTG) in kg. The mothers will be weighed by a scale at the study visit.
Change in adipose tissue mass compared between pregnant women living with HIV and HIV negative pregnant women | <18 weeks (baseline), 32-34 weeks
  Comparison of percent adipose tissue mass per week between pregnant women living with HIV and HIV negative pregnant women during pregnancy.
Change in adipose tissue mass compared between iDTG and cDTG mothers | <18 weeks (baseline), 32-34 weeks
  Comparison of percent adipose tissue mass per week between pregnant women initiating DTG during pregnancy (iDTG) and pregnant women continuing DTG during pregnancy (cDTG).
Differences in maternal metabolic health post-partum between mothers living with HIV and HIV negative mothers | <18 weeks antenatal, 24 weeks postpartum, and 24 months postpartum
  Adiposity will be measured as the main indicator of metabolic health. This outcome focuses on the comparison between mothers living with HIV and HIV negative mothers during pregnancy. Differences in adipose accrual and/or retention will calculated as the difference in adipose (% per week) between the timepoint in question and baseline.
Differences in maternal metabolic health post-partum between iDTG and cDTG mothers | <18 weeks antenatal, 24 weeks postpartum, and 24 months postpartum
  Adiposity will be measured as the main indicator of metabolic health. This outcome focuses on the comparison between mothers initiating DTG during pregnancy and mothers continuing DTG during pregnancy. Differences in adipose accrual and/or retention will calculated as the difference in adipose (% per week) between the timepoint in question and baseline.
Changes in adiposity in the child between HIV positive mothers and HIV negative mothers | <2 weeks, up to 2 years of age
  Adiposity will be measured as the main indicator of metabolic health. This outcome focuses on the comparison between children whose mothers are HIV positive and those whose mothers are HIV negative. Differences in adipose accrual and/or retention will calculated as the difference in adipose (% per week) between the timepoint in question and baseline.
Changes in adiposity in the child between iDTG and cDTG mothers | <2 weeks, up to 2 years of age
  Adiposity will be measured as the main indicator of metabolic health. This outcome focuses on the comparison between children whose mothers initiated DTG during pregnancy and those whose mothers continued DTG during pregnancy. Differences in adipose accrual and/or retention will calculated as the difference in adipose (% per week) between the timepoint in question and baseline.

SECONDARY OUTCOMES:
Changes in subcutaneous adipose tissue (SAT) function | <18 weeks (baseline), 32-34 weeks antenatal, 24 months postpartum
  The SAT sample will reveal information regarding adipocyte hypertrophy, hypoxia, increased fibrosis and inflammation, decreased SAT mitochondrial respiration, and any altered metabolome/lipidome.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine J. Abrams, MD, Principal Investigator — ICAP at Columbia University; Jennifer Jao, MD, Principal Investigator — Northwestern University
Locations (2):
- South Africa (2):
  - Gugulethu Community Health Center, Cape Town
  - Mitchell's Plain Community Health Center, Cape Town

IPD SHARING:
Plan to Share IPD: Yes
As required by study funder, de-identified, archived data will be transmitted to and stored at National Institute of Child Health and Human Development (NICHD)'s Data and Specimen Hub (DASH) for use by other researchers including those outside of the study. Permission to transmit data to DASH will be included in the informed consent signed by all study participants. This data will be shared after the end of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified datasets will be available in DASH no later than 3 years after the completion of baseline study visits.
Access Criteria: When the study is completed, access to study data will be provided through NICHD's DASH repository. Researchers seeking to access data stored in DASH will need to follow pre-specified requirements around data access requests.
URL: http://dash.nichd.nih.gov/